CLINICAL TRIAL: NCT02320318
Title: A 12-week Double-blind, Randomised, Placebo-controlled, Parallel Group Phase III Study, Followed by a 4-week Randomised Withdrawal Period to Evaluate the Efficacy and Safety of Oral Ibodutant 10 mg Once Daily in Female Patients With Irritable Bowel Syndrome With Diarrhoea (IBS-D).
Brief Title: 12-Week Efficacy and Safety Study of Ibodutant in Women With Irritable Bowel Syndrome With Diarrhea (IBS-D)
Acronym: IRIS-05
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAK-08
Record Dates: First submitted 2014-12-12; First posted 2014-12-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Irritable Bowel Syndrome With Diarrhea
Keywords: Irritable Bowel Syndrome; Colon, irritable; Bowel disease; Diarrhea
MeSH Terms: conditions — Irritable Bowel Syndrome; Intestinal Diseases; Diarrhea | interventions — ibodutant; 6-methylbenzo(b)thiophene-2-carboxylic acid (1-(2-phenyl-((1-(tetrahydropyran-4-ylmethyl)piperidin-4-ylmethyl)carbamoyl)ethylcarbamoyl)cyclophenyl)amide; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ibodutant 10 mg (Experimental): Oral tablet once daily for 12 weeks of treatment. At week 13, patients in the ibodutant 10 mg arm will be re-randomised in a 1:1 ratio to either ibodutant 10 mg or placebo for additional 4 weeks of treatment.
  Interventions: Drug: Ibodutant 10 mg
- Placebo (Placebo Comparator): Oral tablet once daily for 12 weeks of treatment. At week 13, patients in the placebo arm will be mock-re-randomised (switch in blinded conditions) to ibodutant 10 mg for additional 4 weeks of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibodutant 10 mg — Oral tablet, once daily.
  Other Names: MEN 15596
  Arms: Ibodutant 10 mg
Drug: Placebo — Oral tablet (identical in appearance and weight to ibodutant tablet), once daily.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome with diarrhoea (IBS-D) is a functional gastrointestinal disorder characterised by chronic or recurrent abdominal pain or discomfort and diarrhoea. The aim of this trial is the evaluation of the efficacy and safety of oral ibodutant 10 mg once daily as compared to placebo in women with IBS-D over a 12-week treatment period.

DETAILED DESCRIPTION:
The study evaluates the efficacy and safety of ibodutant 10 mg, given once daily for 12 weeks in comparison with placebo in female IBS-D patients. Randomisation to ibodutant and placebo will be 1:1. Efficacy is evaluated in terms of weekly response for abdominal pain intensity and stool consistency over 12 weeks of treatment in at least 50% of the weeks of treatment.

The clinical phase of the study comprises up to 2 weeks of screening for patient's eligibility, a 2-week run-in period (treatment-free) for IBS severity assessment, a 12-week double-blind treatment period, a 4-week randomised withdrawal (RW) period and a 2-week safety follow-up, resulting in a maximum 22-week overall duration of the study for each patient.

Patients report their IBS-related symptoms daily in a telephone-based electronic diary from run-in until end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18 years or older.
* Belonging to the Asian race and specifically to the Chinese, Indian and Korean ethnicity.
* Clinical diagnosis of IBS-D according to the following symptoms, based on Rome III modular questionnaire criteria:

  1. Recurrent abdominal pain or discomfort for at least 3 days per month in the last 3 months associated with at least 2 of the following characteristics:

     * improvement with defecation
     * onset associated with a change in the frequency of stool
     * onset associated with a change in form (appearance) of stool.
  2. Symptom-onset at least 6 months prior to diagnosis.
  3. Loose or watery stools at least 25% of the time in the last 3 months AND hard or lumpy stools less than 25% of the time in the last 3 months.
  4. Additional criterion: More than 3 bowel movements per day at least 25% of the time in the last 3 months.
* For patients older than 50 years OR patients with a positive family history of colorectal cancer: Normal results from colonoscopy/flexible sigmoidoscopy performed within the last 5 years.
* For patients aged 65 years or older: Absence of ischaemic colitis, microscopy colitis or any other organic gastrointestinal disease as evidenced by the results of a colonoscopy/flexible sigmoidoscopy with biopsy performed within 6 months.
* For women of childbearing potential: Use of a highly effective contraceptive method with a failure rate <1% per year throughout the entire study period.
* Physical examination without clinically relevant abnormalities during screening.
* No clinically relevant abnormalities in 12-Lead ECG or in laboratory findings.
* Mentally competent, able to give written informed consent, and compliant to undergo all visits and procedures.
* Unrestricted access to a touch-tone telephone.
* Willingness to refrain from using loperamide within 3 days prior to run-in visit and during the run-in period.

Additional criteria at randomisation:

* During both weeks of the run-in period:

  1. A weekly average of worst abdominal pain in the past 24 hours with a score of ≥3.0 on a 0 to 10 point scale.
  2. At least one bowel movement on each day.
  3. A weekly average of at least 3 bowel movements per day.
  4. At least one stool with a consistency of Type 6 or Type 7 according to the Bristol Stool Scale (BSS) on at least 2 days per week.
  5. Less than 2 bowel movements with a consistency of Type 1 or Type 2 according to the BSS per week.
* Adequate compliance with the e-diary recording procedure defined as at least 11 of 14 days (≥75%) of the nominal daily data entry.

Exclusion Criteria:

* Male gender.
* Diagnosis of IBS with a subtype of constipation, mixed IBS, or un-subtyped IBS.
* Colonic or major abdominal surgery, any other major abdominal surgery or elective major surgery planned or expected during the study.
* History of organic GI abnormalities, inflammatory bowel diseases, complicated diverticulosis, ischaemic colitis, microscopic colitis.
* History of pancreatitis, active biliary duct disease, cholecystitis or symptomatic gallbladder stone disease in the previous 6 months.
* History of gluten enteropathy or lactose intolerance.
* Current or previous diagnosis of neoplasia.
* History of endometriosis.
* History of positive tests for ova or parasites, or clostridium difficile toxin or occult blood in the stool in the previous 6 months.
* History of human immunodeficiency virus infection.
* History of major cardiovascular events in the previous 6 months.
* Uncontrolled hypertension, insulin-dependent diabetes mellitus or abnormal thyroid function.
* Major psychiatric or neurological disorders or unstable medical condition which may compromise the efficacy and safety assessments.
* Evidence of clinically significant hepatic disease, severe renal insufficiency or anemia.
* Relevant changes in dietary habits, lifestyle, or exercise regimen in the previous 2 months.
* Use of prohibited concomitant medication within the previous month such as antibiotics, antimuscarinic drugs, drugs enhancing GI motility and analgesics.
* Pregnancy or breastfeeding.
* Inability to understand or collaborate throughout the study.
* Participation in other clinical studies in the previous 4 weeks or concomitant enrollment in a clinical study.
* Any condition that would compromise the well-being of the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Weekly response for abdominal pain intensity AND stool consistency over 12 weeks of treatment in at least 50% of the weeks of treatment (6 out of 12 weeks). | 12-week
  The patient will be considered a weekly responder if she meets both of the following criteria in the same week:
  * Abdominal pain response: decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline;
  * Stool consistency response: decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.

SECONDARY OUTCOMES:
Weekly response for abdominal pain intensity over 12 weeks of treatment in at least 50% of the weeks of treatment (6 out of 12 weeks). | 12-week
  The patient will be considered a weekly abdominal pain responder if she meets the following criterion:
  * Decrease in weekly average of worst abdominal pain score in the past 24 hours of at least 30% compared with baseline.
Weekly response for stool consistency over 12 weeks of treatment in at least 50% of the weeks of treatment (6 out of 12 weeks). | 12-week
  The patient will be considered a weekly stool consistency responder is she meets the following criterion:
  * Decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline.
Weekly Response for relief of overall IBS signs and symptoms over 12 weeks of treatment in at least 50% of the weeks of treatment (6 out of 12 weeks). | 12-week
  The patient will be considered a weekly responder if she has an IBS degree-of-relief equal to "completely relieved/improved" or "considerably relieved/improved".
Evaluation of rebound effects | 12-week
  Comparison between average abdominal pain intensity and stool consistency during the 4-week RW treatment period and baseline in patients who are re-randomised to placebo after being treated with ibodutant.

CONTACTS AND LOCATIONS:
Overall Officials: Jan F Tack, Prof., Study Chair — Department of Gastroenterology, University Hospital Gasthuisberg, Katholieke Universiteit Leuven, Leuven, Belgium
Locations (12):
- Singapore, Singapore
- South Korea (5):
  - Busan
  - Daegu
  - Gangwon-do
  - Gyeonggi-do
  - Seoul
- Taiwan (6):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan District
  - Yunlin